CLINICAL TRIAL: NCT02775786
Title: Assessing the Utility of Macromolecular Dynamic Contrast Enhanced MRI and Diffusion Weighted Imaging as Biomarkers for Vascular Permeability and Fibrosis in Pancreatic Cancer
Brief Title: Prospective Evaluation of MRI Biomarkers in Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAL2505
Record Dates: First submitted 2015-02-25; First posted 2016-05-18 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic Adenocarcinoma; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (No Intervention): Normal volunteers with no pancreas mass or risk factors for pancreas cancer will be recruited for MRI protocol optimization and nothing more. No intravenous contrast will be given. They will be asked to lie in the scanner for up to 1 hour and non-contrast imaging will be performed.
- Pancreatic Mass or Risk Factors Group (Experimental): Participants with pancreatic adenocarcinoma who are planning to undergo surgical resection. Participants will undergo up to two MRIs with and without intravenous contrast. The first MRI will be performed using an extracellular contrast agent and the second 1-14 days later, with a macromolecular contrast agent. If patient cannot undergo the second MRI for any reason eg. not enough time before surgery, one MRI with either contrast agent will still be used for analysis .
  Interventions: Other: MRIs with and without intravenous contrast (up to 2)

INTERVENTIONS:
Other: MRIs with and without intravenous contrast (up to 2) — Participants will undergo up to two MRIs with and without intravenous contrast. The first MRI will be performed using an extracellular contrast agent and the second 1-14 days later, with a macromolecular contrast agent. If patient cannot undergo the second MRI for any reason eg. not enough time before surgery, one MRI with either contrast agent will still be used for analysis.
  Arms: Pancreatic Mass or Risk Factors Group

SUMMARY:
This is a prospective cohort study in participants with pancreatic adenocarcinoma who are undergoing surgical resection. Participants will have up to two magnetic resonance imaging (MRI) scans with and without intravenous contrast. The MRI will be performed using either an extracellular contrast agent or using a macromolecular contrast agent. These contrast agents are routinely used in body MRI and are on formulary at this institution. Parameters will be compared to histopathology measures of mean vascular density and grade of fibrosis, respectively. The purpose is to establish a standard protocol for future clinical trials of treatments that would use MRI parameters as quantitative markers of treatment effect.

DETAILED DESCRIPTION:
This is a prospective cohort study of dynamic contrast enhanced MRI (DCE-MRI), which includes diffusion weighted imaging (DWI-MRI) in participants with pancreatic adenocarcinoma who are undergoing surgical resection. Participants will have up to two MRI scans with and without intravenous contrast. The MRI will be performed using either an extracellular contrast agent or using a macromolecular contrast agent. These contrast agents are routinely used in body MRI and are on formulary at this institution. Quantitative parameters of volume transfer coefficient (Ktrans) and apparent diffusion coefficient (ADC) will be calculated from the MRI sequences and each parameter will be compared to histopathology measures of mean vascular density and grade of fibrosis, respectively. The influence of the contrast agent (extracellular and macromolecular) on agreement between imaging parameters and histopathology will be assessed and agreement in Ktrans as derived from a one compartment and a two-compartment model will be assessed. If a participant is unable to receive intravenous contrast due to renal dysfunction or refuses IV contrast, the non-contrast portion of the exam will be used for analysis. The purpose is to establish a standard protocol for future clinical trials of treatments that would use MRI parameters as quantitative markers of treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age.
2. Biopsy proved pancreatic ductal adenocarcinoma (PDA) and/or a pancreatic mass with imaging features suggestive of pancreatic adenocarcinoma planned for surgical resection.
3. No contraindication to MRI such as severe claustrophobia (not alleviated by oral anti-anxiolytics) or metal/mechanical devices in their body not considered magnetic resonance (MR) compatible at 1.5 Tesla (departmental MRI safety screening form)
4. No known allergy to gadolinium based contrast agent
5. For contrast enhanced studies, participant has an estimated glomerular filtration rate (GFR) >30 mg/dL using the modification of diet in Renal Disease (MDRD) formula. If the participant has an estimated GFR ≤30 mg/dL, they can still participate but no intravenous contrast will be administered.

Exclusion Criteria:

1. Contraindication to MR imaging
2. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Correlation between Apparent Diffusion Coefficient (ADC) of pancreatic cancer based on MRI with percent fibrosis at histopathology | One year

SECONDARY OUTCOMES:
Correlation between Ktrans of pancreatic cancer derived from dynamic contrast enhanced MRI performed with gadopentetate dimeglumine and mean vascular density quantified at histopathology. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Luk, MD, Principal Investigator — CUIMC
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided